CLINICAL TRIAL: NCT02446769
Title: A Pilot, Multi-Center, Randomized, Open-Label, Parallel Group Study to Assess the Effects of a Novel Application of Averaged Volume Assured Pressure Support Ventilation (AVAPS-AE) Therapy on Re-hospitalization in Patients With Sleep-Disordered Breathing With Co-morbid COPD
Brief Title: A Pilot Study to Assess the Effects of a Novel Application of Averaged Volume Assured Pressure Support Ventilation (AVAPS-AE) Therapy on Re-hospitalization in Patients With Sleep-Disordered Breathing With Co-morbid COPD
Acronym: STOP-BBACK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting patient population.
Sponsor: Philips Respironics (Industry)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRC-1426-BBACK-MS
Record Dates: First submitted 2015-04-09; First posted 2015-05-18 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Breathing-Related Sleep Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AVAPS-AE Non-invasive ventilation therapy (Experimental): Participants will be initiated on AVAPS-AE therapy (intervention arm) for 60 days. AVAPS-AE is a mode of therapy (Philips Respironics Inc, Monroeville, Pa) with potential advantages over the currently established modes of non-invasive positive pressure ventilation (CPAP and bilevel therapy). This mode of therapy incorporates AVAPS (automated adjustable Inspiratory Positive Airway Pressure (IPAP) setting to maintain target ventilation with a settable rate of change), Auto Expiratory Positive Airway Pressure (EPAP) and Auto Back up Rate.
  Interventions: Device: AVAPS-AE Non-invasive ventilation therapy
- Standard of Care Group (No Intervention): Evaluation and treatment of the participant's sleep disordered breathing will be per their participant's health care provider's usual care pathway.

INTERVENTIONS:
Device: AVAPS-AE Non-invasive ventilation therapy — Participants will use the device greater than or equal to 4hrs per night for the 60 days after discharge.
  Arms: AVAPS-AE Non-invasive ventilation therapy

SUMMARY:
This is a multicenter, randomized, parallel-group, open label study of the efficacy of AVAPS-AE to prevent re-hospitalization in hospitalized patients with comorbid Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
This is a multicenter, randomized, parallel-group, open label study of the efficacy of AVAPS-AE to prevent re-hospitalization in hospitalized patients with comorbid COPD. Hospitalized patients with comorbid COPD who are at high risk for readmission will be recruited. Specifically patients with comorbid COPD who are to be discharged with (a) admission diagnosis of COPD (GOLD stage II or greater); AND (b) either a prior non-elective hospitalization (one in the past 12 months) OR active smoker. Such participants will undergo questionnaire-based screening for sleep-disordered breathing (STOP-BANG questionnaire) and if they have a high risk for Sleep Disordered Breathing (SDB) (> 3 points) will undergo an overnight portable sleep study for screening prior to hospital discharge (AHI > 10 per hour; >3% oxygen desaturation for hypopneas).

After randomization and prior to discharge, participants will either be initiated on AVAPS-AE therapy (intervention arm) for 60 days or will be referred to the sleep center for further diagnostic testing and therapy initiation (standard of care arm). Participants will complete quality of life questionnaires Functional outcomes of sleep questionnaire (FOSQ) at baseline (in-person), and in 30 and 60 days (by mail) post discharge. Information regarding hospital admission, diagnostic tests, medication changes, and procedures will be collected from all participants. Discharge summaries of re-hospitalizations and office or ER visits, as well as diagnostics tests and therapies received will be collected for measuring healthcare costs.

Participants will have an option to enroll in a registry for a 3 year follow-up and will also be queried on a yearly basis regarding hospitalizations, cardiovascular events, and assessment of vital statistics in the National Death Index registry. The study will conclude when all randomized participants have been followed for a minimum of 60 days.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients who are at high risk for readmission who are at least 18 years of age.
2. Specifically patients with (a) admission diagnosis of COPD AND (b) either a prior non-elective hospitalization (One in the past 12 months) OR active smoker who are ready for discharge AND (c) are also found to have sleep-disordered breathing (AHI ≥ 10 per hour; >3% oxygen desaturation for hypopneas) by overnight portable respiratory study prior to hospital discharge.
3. Bedside spirometry revealing evidence for obstructive lung disease (post-bronchodilator; GOLD stage II or greater (FEV1 <70% predicted post BD).
4. No previous home Positive Airway Pressure (PAP) or Non- Invasive Ventilation (NIV) use within the past year

Exclusion Criteria:

1. Central sleep apnea (Central apnea index >5 per hour; and/or >50% are central apneas & hypopneas)
2. Clinically unstable, i.e., Acute Respiratory Failure, hypotensive shock, uncontrolled cardiac ischemia or arrhythmias, requiring life support ventilation or as otherwise determined by the investigator
3. Participants with Stage III & IV Chronic Heart Failure as defined by the New York Heart Association (NYHA) Classification
4. Known or expected contraindications for the use of non-invasive ventilation per the assessment of the investigator.
5. Lack of medical insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sairam Parthasarathy, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Background] Briones Claudett KH, Briones Claudett M, Chung Sang Wong M, Nuques Martinez A, Soto Espinoza R, Montalvo M, Esquinas Rodriguez A, Gonzalez Diaz G, Grunauer Andrade M. Noninvasive mechanical ventilation with average volume assured pressure support (AVAPS) in patients with chronic obstructive pulmonary disease and hypercapnic encephalopathy. BMC Pulm Med. 2013 Mar 12;13:12. doi: 10.1186/1471-2466-13-12. PMID 23497021
- [Background] Marin JM, Soriano JB, Carrizo SJ, Boldova A, Celli BR. Outcomes in patients with chronic obstructive pulmonary disease and obstructive sleep apnea: the overlap syndrome. Am J Respir Crit Care Med. 2010 Aug 1;182(3):325-31. doi: 10.1164/rccm.200912-1869OC. Epub 2010 Apr 8. PMID 20378728
- [Background] Jencks SF, Williams MV, Coleman EA. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Apr 2;360(14):1418-28. doi: 10.1056/NEJMsa0803563. PMID 19339721
- [Background] Westert GP, Lagoe RJ, Keskimaki I, Leyland A, Murphy M. An international study of hospital readmissions and related utilization in Europe and the USA. Health Policy. 2002 Sep;61(3):269-78. doi: 10.1016/s0168-8510(01)00236-6. PMID 12098520

RESULTS

PARTICIPANT FLOW:
Groups:
- Screening Period: All participants that signed the consent.
- Standard of Care: Evaluation and treatment of the participant's sleep disordered breathing will be per their participant's health care provider's usual care pathway.
- Experimental: AVAPS-AE Non-invasive Ventilation Therapy: Participants will be initiated on AVAPS-AE therapy (intervention arm) for 60 days. AVAPS-AE is a mode of therapy (Philips Respironics Inc, Monroeville, Pa) with potential advantages over the currently established modes of non-invasive positive pressure ventilation (CPAP and bilevel therapy). This mode of therapy incorporates AVAPS (automated adjustable Inspiratory Positive Airway Pressure (IPAP) setting to maintain target ventilation with a settable rate of change), Auto Expiratory Positive Airway Pressure (EPAP) and Auto Back up Rate.
Period: Screening Period
Arm/Group | Screening Period | Standard of Care | Experimental: AVAPS-AE Non-invasive Ventilation Therapy
Started | 18 | 0 | 0
Completed | 7 | 0 | 0
Not Completed | 11 | 0 | 0
Not completed — Screen Failure | 11 | 0 | 0
Period: Study Period
Arm/Group | Screening Period | Standard of Care | Experimental: AVAPS-AE Non-invasive Ventilation Therapy
Started | 0 | 4 | 3
Completed | 0 | 2 | 3
Not Completed | 0 | 2 | 0
Not completed — Randomized in Error | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Due to the low enrollment, and low number of participants randomized into the study baseline analysis population description data was combined to provide more purposeful data.
Groups:
- All Participants: All participants that were consented.
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 18
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 39 (8.17)
Current Smokers [Count of Participants; unit: Participants] | 7
Gold Stage [Count of Participants; unit: Participants] — GOLD is the Global Initiative for Chronic Obstructive Lung Disease stage or grade. Doctors assign grades based on four separate pieces of information:
  How severe your current symptoms are, your spirometry results,the chances that your COPD will get worse, and the presence of other health problems. The higher the stage the more severe the COPD.
  Participants
    Gold Stage II | 4
    Gold Stage III | 4
    Gold Stage IIII | 1
    Unknown | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Enrolled Requiring Emergent Healthcare (Such as Re-hospitalization, Unscheduled Physician Office Visits, Urgent Care Visits or Emergency Room Visits).
Description: Evaluate the effects of novel application of Averaged Volume Assured Pressure Support (AVAPS-AE) therapy on the number of participants with emergent and non-emergent healthcare utilization with sleep-disordered breathing who are hospitalized with co-morbid Chronic Obstructive Pulmonary Disease (COPD), number of participants enrolled.
Time Frame: 60 days post-discharge
Measure: Count of Participants; unit: Participants
Groups:
- AVAPS-AE Non-invasive Ventilation Therapy: Participants will be initiated on AVAPS-AE therapy (intervention arm) for 60 days. AVAPS-AE is a mode of therapy (Philips Respironics Inc, Monroeville, Pa) with potential advantages over the currently established modes of non-invasive positive pressure ventilation (CPAP and bilevel therapy). This mode of therapy incorporates AVAPS (automated adjustable IPAP setting to maintain target ventilation with a settable rate of change), Auto EPAP and Auto Back up Rate.
  AVAPS-AE Non-invasive ventilation therapy: Participants will use the device greater than or equal to 4hrs per night for the 60 days after discharge.
Arm/Group | AVAPS-AE Non-invasive Ventilation Therapy | Standard of Care Group
Number analyzed (Participants) | 3 | 2
Participants | 1 | 0

2. Primary Outcome: Composite End-point of Time (# of Days) to Occurrence of Emergent Healthcare Utilization (Such as Re-hospitalization, Unscheduled Physician Office Visits, Urgent Care Visits or Emergency Room Visits).
Description: Evaluate the effects of novel application of Averaged Volume Assured Pressure Support (AVAPS-AE) therapy on time to (# of days) emergent and non-emergent healthcare utilization in patients with sleep-disordered breathing who are hospitalized with co-morbid Chronic Obstructive Pulmonary Disease (COPD).
Time Frame: 60 days post-discharge
Population: Only one participant enrolled in the study required emergent healthcare utilization.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AVAPS-AE Non-invasive Ventilation Therapy | Standard of Care Group
Number analyzed (Participants) | 1 | 0
days | 21 (0) |

3. Secondary Outcome: Healthcare Costs
Description: Evaluate the effects of novel application of Averaged Volume Assured Pressure Support (AVAPS-AE) therapy on the number of emergent and non-emergent healthcare utilization over 6 months; costs related to re-hospitalization; number of visits to physician offices or emergency rooms, and health-related quality of life (disease-specific and general HR-QOL measures).
Time Frame: 60 days post-discharge
Population: Data was not collected as study was terminated.
Arm/Group | AVAPS-AE Non-invasive Ventilation Therapy | Standard of Care Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Quality of Life (SF-36) at 30 and 60 Days
Description: Evaluate the effects of novel application of Averaged Volume Assured Pressure Support (AVAPS-AE) therapy on health-related quality of life. The Short Form 36 (SF-36) is a set of quality of life measures. Participants were asked at 30 days and 60 days in general what their overall health was. On a scale of 1 to 5 -1 being excellent, 5 being poor.
Time Frame: 30 and 60 days post-discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVAPS-AE Non-invasive Ventilation Therapy | Standard of Care Group
Number analyzed (Participants) | 3 | 2
units on a scale
  30 days | 3.3 (1.41) | 4 (0)
  60 days | 3.7 (3.5) | 3.5 (0.7)

5. Secondary Outcome: Change in Quality of Life (FOSQ) at 30 and 60 Days
Description: FOSQ is a quality of life questionnaire for sleep disorders. It's a 30 question survey with 5 subgroups: general productivity (8 questions), social outcome (2 questions),activity level (9 questions), vigilance (7 questions) and intimate relationships & sexual activity (4 questions).
  Scores are provided on a 0 to 4 scale:
  0- I don't do this activity for other reasons or missing response
  1- Yes, extreme difficulty 4- no difficulty The average score was calculated based upon average sub-scores. The total score was, calculated using the mean of the subscale scores and multiplying the mean by the number of subscales. The range of scores for the total score is 5-20. The measures are designed to assess the impact of disorders of excessive sleepiness on activities of everyday living and the extent to which these abilities are improved by effective treatment. The lower the score the more difficulty a person has carrying out certain activities because they are too sleepy or tired.
Time Frame: 30 and 60 days post-discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVAPS-AE Non-invasive Ventilation Therapy | Standard of Care Group
Number analyzed (Participants) | 3 | 2
units on a scale
  30 Days | 15.1 (6.6) | 18.8 (0)
  60 Days | 15.5 (4.3) | 19.3 (0.5)

6. Secondary Outcome: Composite End-point of Time to Occurrence of Non-emergent Healthcare Utilization (Such as Scheduled Hospitalization, Scheduled Physician Office, Urgent Care Visits or Emergency Room Visits).
Description: as for outcome 3
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AVAPS-AE Non-invasive Ventilation Therapy | Standard of Care Group
Number analyzed (Participants) | 3 | 2
days | 0 (0) | 0 (0)

7. Secondary Outcome: Time to Re-hospitalization Alone
Description: Evaluate the effects of novel application of Averaged Volume Assured Pressure Support (AVAPS-AE) therapy on time to re-hospitalization alone.
Time Frame: 60 days post-discharge
Population: Only one enrolled participation was hospitalized.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AVAPS-AE Non-invasive Ventilation Therapy | Standard of Care Group
Number analyzed (Participants) | 1 | 0
days | 21 (0) |

8. Secondary Outcome: Number of Hospitalizations Over 3 Years (Optional if Enrolled in Registry)
Description: as for outcome 3
Time Frame: 3 years
Population: No participants were enrolled in the registry.
Arm/Group | AVAPS-AE Non-invasive Ventilation Therapy | Standard of Care Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 days
Groups:
- Experimental: AVAPS-AE Non-invasive Ventilation Therapy: Participants will be initiated on AVAPS-AE therapy (intervention arm) for 60 days. AVAPS-AE is a mode of therapy (Philips Respironics Inc, Monroeville, Pa) with potential advantages over the currently established modes of non-invasive positive pressure ventilation (CPAP and bilevel therapy). This mode of therapy incorporates AVAPS (automated adjustable IPAP setting to maintain target ventilation with a settable rate of change), Auto EPAP and Auto Back up Rate.
Arm/Group | Screening Period | Standard of Care | Experimental: AVAPS-AE Non-invasive Ventilation Therapy
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/4 | 1/3
Other Adverse Events (participants affected / at risk) | 0/18 | 0/4 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening Period (N=18) | Standard of Care (N=4) | Experimental: AVAPS-AE Non-invasive Ventilation Therapy (N=3)
Hyperkalemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Cardiac Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Fall secondary loss of consciousness (General disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was terminated early due to a high number of screen failures therefore data analysis with any statistical significance could not be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT02446769/Prot_SAP_000.pdf